CLINICAL TRIAL: NCT01320787
Title: A Phase I Study of 18-F-Fluoroacetate Sodium as a PET Imaging Agent for Tumor Detection
Brief Title: 18-F-Fluoroacetate as PET Imaging Agent
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-0157; NCI-2011-01066 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Brain Cancer; Breast Cancer; Prostate Cancer
Keywords: Brain; Adenocarcinoma of the prostate; Locally advanced breast cancer; Estrogen receptor; ER; Progesterone receptor; PR; Negative for ErbB2; Malignant tumor of the central nervous system; CNS
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Central Nervous System Neoplasms | interventions — fluoroacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-fluoroacetate (Experimental): 18F-fluoroacetate injection as a single intravenous bolus with a maximum volume of 4 mL followed by a saline flush of 20 to 50 mL.
  Interventions: Drug: 18F-fluoroacetate

INTERVENTIONS:
Drug: 18F-fluoroacetate — 18F-fluoroacetate injection as a single intravenous bolus with a maximum volume of 4 mL followed by a saline flush of 20 to 50 mL.

SUMMARY:
The goal of this clinical research study is to find out the highest tolerable dose of an imaging solution called 18-F-fluoroacetate sodium that can be given before a positron emission tomography (PET) scan. The safety of this solution will also be studied.

DETAILED DESCRIPTION:
The Study Solution:

18-F-fluoroacetate sodium is designed to be attracted to cells that grow in some tumors. This imaging solution has a small dose of radiation added to it, which may help the doctor to "see" cancer cells and their possible spread through the body, during the scans. This is the first study using 18-F-fluoroacetate sodium in humans.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to an imaging study date. The first group of 6 participants will receive a smaller dose of solution (less than one half of the regular PET scan tracer radioactivity). The later 2 groups may receive the same dose of solution or a larger dose, but the larger dose will still be no more than what you would receive in a regular clinic PET scan procedure.

Study Solution Administration and PET Scans:

On Day 1, you will receive 18-F-fluoroacetate sodium by vein over 5 minutes.

You will then have 3 PET scans with a PET/CT scanner. You will be lying down during the PET scan. Each scanning period will take about 1 hour. You will have a 20-minute rest period between each scan.

Before each PET scan, you will have a CT scan, called a "Scout View", to check your position in the machine. This should take about 5 minutes.

You may continue receiving standard treatment from your regular doctor throughout the entire time you are in this study.

Study Visits:

On Day 1 (the day of the injection and imaging study):

* You will have an ECG, your vital signs will be measured, and the injection site will be checked at 5 minutes before, and 30 minutes and 2 ½ hours after the imaging solution is injected.
* You will be asked if you have had any side effects.
* Blood (about 2 tablespoons total) will be drawn 9 times over 2 ½ hours after the injection for pharmacokinetic (PK) testing. PK testing measures the amount of the imaging solution in the body at different time points.
* Urine will also be collected to test the amount of radiation that might have been absorbed by the body. This will be collected during the 10 minute rest periods.

On Day 2:

* Your vital signs will be measured.
* You will have an ECG.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* The injection site will be checked.
* You will be asked if you have had any side effects.

On Day 7:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* The injection site will be checked.
* You will be asked if you have had any side effects.

On about Day 30:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* The injection site will be checked.
* You will be asked if you have had any side effects.

Length of Study:

You will be on active study for the day you receive the imaging and 18-F-fluoroacetate sodium. You will be on follow-up for up to 30 days after the imaging.

This is an investigational study. 18-F-fluoroacetate sodium is not FDA approved or commercially available. At this time, it is being used in research only. The study scans are also considered investigational when used for this purpose, and will not be used for planning your cancer treatment.

Up to 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have: a) Histologic or cytologic confirmation of adenocarcinoma of the prostate; or b) A histologically confirmed, treatment-naïve, locally advanced breast cancer that express either estrogen receptor (ER) or progesterone receptor (PR) and are negative for ErbB2 by Immunohistochemistry (IHC) and/or fluorescence in situ hybridization (FISH) gene amplification; or c) Suspected supratentorial malignant primary or secondary malignant tumor of the central nervous system (CNS).
2. The Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2 or Karnofsky Performance Status of ≥ 60.
3. Four weeks or greater since major surgery.
4. Required Initial Laboratory Data: a) White Blood Count (WBC) >/= 3,000/microliters. b) Absolute neutrophil count (ANC) >/= 1,500/microliters. c) Platelet count >/= 100,000/microliters. d) Creatinine </= 1.5 x upper limit of normal e) Bilirubin </= 2 x upper limit of normal (exceptions will be made for patients with Gilbert's Disease). f) SGOT (AST) </= 2.5 x upper limit of normal. g) SGPT (ALT) </= 2.5 x upper limit of normal.
5. Subjects must be at least 18 years of age
6. All sexually active subjects of child-bearing potential (CBP) must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of study participation from signing of consent till 30 days post injection. Should a male patient's sexual partner become pregnant or suspects that she is pregnant while the patient is participating in the study, the treating physician should be notified immediately. Female subjects of CBP must have a negative serum pregnancy test within 24 hours prior to the administration of the protocol imaging agent.
7. For patients with adenocarcinoma of the prostate, they must have radiographic evidence of metastatic prostate cancer; measurable lymph node disease on either CT scan, MRI with any level of serum PSA. (There is no limitation of the type or numbers of prior chemotherapy regimens, palliative radiotherapy or other non-chemotherapy or hormonal therapies for metastatic disease.)
8. For subjects with breast cancer, they must have local disease evaluated by standard breast imaging before initiation of treatment and no evidence of metastatic disease.
9. For subjects with a recent biopsy of newly diagnosed high-grade tumor, they must have recovered from the effects of surgical biopsy. It must be at least >/= 7 days after a brain biopsy to be eligible.
10. Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed imaging agent.
11. Baseline imaging of all tumor types must be within 21 days of protocol PET imaging day, but more than 24 hours prior to the protocol PET imaging tracer administration. Patients can receive other standard diagnostic imaging procedures 24 hours post protocol PET imaging day.

Exclusion Criteria:

1. Patients with significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months) are excluded.
2. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition (i.e. 18F-FDG)
4. Patients may not be receiving any other investigational agents while on this protocol.
5. Patients with prostate cancer may not be receiving dutasteride or finasteride up to 2 weeks prior to enrollment.
6. Patients who have received prior cytotoxic, biologic, hormonal (other than for replacement) therapy to treat the breast cancer. (Patients may continue on a daily Multi-Vitamin and any other herbal, alternative or food supplements.)
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into the study.
8. Patients with metastatic adenocarcinoma of the prostate documented by bone scan alone, are ineligible.
9. Sexually active fertile men not using effective birth control if their partners are women of childbearing potential (WOCBP).
10. Women who are pregnant, not using effective birth control or lactating are ineligible
11. The subject is unable to lie down for 150 minutes.
12. The subject suffers from claustrophobia.
13. The subject has a history of serious hypersensitivity reaction to iodinated contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 18F-Fluoroacetate | 1 day
  Biodistribution of 18F-fluoroacetate is measured during imaging, using a radioisotope (18F) of fluoroacetate PET scan. The percent injected dose (%ID) obtained in different organs derived from the PET data.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Podoloff, MD, BA, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org